CLINICAL TRIAL: NCT06084923
Title: Outcomes of Unfit Patients With Chronic Lymphocytic Leukemia (CLL) Included in the Front-line GIMEMA LLC1114 Trial Who Discontinued Ibrutinib Due to Reasons Other Than Disease Progression: a Multicenter Retrospective/ Prospective Observational Study.
Brief Title: Outcomes of Unfit Patients With CLL Included in the GIMEMA LLC1114 Trial Who Discontinued Ibrutinib Due to Reasons Other Than Disease Progression
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CLL2523
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who discontinued ibrutinib: CLL patients enrolled in the front-line GIMEMA LLC1114 study twho discontinued ibrutinib due to reasons other than CLL progression, Richter syndrome, malignancy or death, or lost to the follow-up.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Patients will be observed after ibrutinib discontinuation and data on ibrutinib discontinuation, reatreatment and outcome will be collected

SUMMARY:
The goal of this observational study is to assess in the cohort of CLL patients enrolled in the front-line GIMEMA LLC1114 study who discontinued ibrutinib the time to subsequent treatment. The main question it aims to answer is:

• The 12 and 24-month TTNT measured from the time of ibrutinib discontinuation due to reasons other than CLL progression, Richter syndrome, malignancy or death, or lost to the follow-up.

Participants will be observed for the duration of the study.

DETAILED DESCRIPTION:
This is an observational, multicenter, retrospective and prospective study aimed at analyzing in the cohort of CLL patients enrolled in the front-line GIMEMA LLC1114 study the time to next treatment in patients who discontinued ibrutinib due to reasons other than CLL progression, Richter syndrome, malignancy or death, or lost to the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with ibrutinib included in the LLC1114 GIMEMA study who have discontinued ibrutinib after completing 78-months of treatment per protocol OR patients treated with ibrutinib included in the LLC1114 GIMEMA study who were treated for at least 12 months before discontinuing ibrutinib due to reasons other than CLL progression, Richter syndrome, malignancy or death, or lost to the follow-up and had achieved a response (CR or PR/PR-L) lasting at least 6 months before discontinuing ibrutinib
* Informed consent, if applicable.

Exclusion Criteria:

- Patients with concomitant conditions that may interfere with an appropriate assessment of the TTNT in the physician opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patients enrolled in the front-line GIMEMA LLC1114 study who discontinued ibrutinib due to reasons other than CLL progression, Richter syndrome, malignancy or death, or lost to the follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The 12 and 24-month Time To Next Treatment (TTNT) measured from the time of ibrutinib discontinuation due to reasons other than CLL progression, Richter syndrome, malignancy or death, or lost to the follow-up. | 12 and 24 months
  The 12 and 24-month time to the next treatment (TTNT) will be calculated in terms of the proportion of patients who requiring new treatment at 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Francresca Romana Mauro, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No